CLINICAL TRIAL: NCT04495764
Title: Registry of Sustained Immunity to COVID-19 Among ESKD Patients
Acronym: RePAiR
Status: Completed | Type: Observational
Sponsor: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-M-0044-00
Record Dates: First submitted 2020-07-22; First posted 2020-08-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: SARS-CoV-2 Infection; Anti-SARS-CoV-2 Infection
Keywords: Immunoglobulin G; Immunoglobulin M
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Baseline serologic characterization for anti-SARS-CoV-2 IgM and IgG
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center, prospective registry study of subjects undergoing hemodialysis for treatment of end-stage renal disease in a DaVita center.

The objective of this study is to understand whether and to what degree anti-SARS-CoV-2 antibodies mitigate the risk of subsequent SARS-CoV-2 infection and COVID disease within the ESKD population.

DETAILED DESCRIPTION:
This is a multi-center, prospective registry study of subjects undergoing hemodialysis for treatment of end-stage renal disease in a DaVita center.

The objective of this study is to understand whether and to what degree anti-SARS-CoV-2 antibodies mitigate the risk of subsequent SARS-CoV-2 infection and COVID disease within the ESKD population.

Following informed consent, participants will undergo baseline serologic characterization for anti-SARS-CoV-2 IgM and IgG. The study is planned to align with the present wave of COVID-19. Enrollment will continue until the total sample size of 2500 is reached or until the study sponsor determines. Should there be a subsequent wave of COVID- 19, participants will be actively surveiled for evidence of SARS-CoV-2 infection and for COVID-19 disease. The relationship between baseline serologic status and subsequent infection/disease will be determined.

This study will have 2 distinct phases.

Phase 1 (baseline characterization) start will be triggered by the sponsor and may start at different times at the active sites. Participants will be consented and enrolled and blood will be collected for anti-SARS-CoV-2 antibodies.

Phase 2: Start will be triggered by the sponsor in the fall of 2020 and each geographic study location may be triggered to start at separate times. Study participants will be followed prospectively for incidence and severity of COVID-19. Study visits will commence upon sponsor trigger and will occur once monthly for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Between ≥18 and 80 years of age, inclusive.
* Ability to provide informed consent.
* Currently receiving hemodialysis treatment for end-stage kidney disease at a DaVita dialysis center.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Between ≥18 and 80 years of age, inclusive.
  2. Ability to provide informed consent.
  3. Currently receiving hemodialysis treatment for end-stage kidney disease at a DaVita dialysis center.
Sampling Method: Non-Probability Sample
Enrollment: 2315 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 antibodies | Through study completion (5 visits), an average of 6 months
Incidence and severity of COVID-19 | Through study completion (5 visits), an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Tentori, MD, Principal Investigator — Davita Clinical Research
Locations (11):
- United States (11):
  - DCR Victorville, Victorville, California
  - DCR Connecticut, Bridgeport, Connecticut
  - DCR Twin Cities, Minneapolis, Minnesota
  - DCR Las Vegas, Las Vegas, Nevada
  - DCR Bronx, The Bronx, New York
  - DCR Canton, Canton, Ohio
  - DCR El Paso, El Paso, Texas
  - DCR Lewisville, Lewisville, Texas
  - DCR San Antonio, San Antonio, Texas
  - DCR Norfolk, Norfolk, Virginia
  - DCR Milwaukee, Milwaukee, Wisconsin